CLINICAL TRIAL: NCT04701372
Title: Clinical Outcomes From NOCD Digital Behavioral Health Treatment of Obsessive-Compulsive Disorder Using Exposure and Response Prevention
Brief Title: Clinical Outcomes From NOCD Treatment of Obsessive-Compulsive Disorder Using Exposure and Response Prevention
Status: Completed | Type: Observational
Sponsor: NOCD (Industry)
Responsible Party: Sponsor
Other Study IDs: NOCD001
Record Dates: First submitted 2021-01-02; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: exposure and response prevention; digital behavioral health; remote treatment; video therapy
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obsessive-Compulsive Disorder: adults, adolescents, and children with obsessive-compulsive disorder
  Interventions: Behavioral: Exposure and response prevention therapy

INTERVENTIONS:
Behavioral: Exposure and response prevention therapy — Exposures and response prevention therapy (a type of cognitive-behavioral therapy for obsessive-compulsive disorder), delivered in real-time by licensed therapists remotely via video. The treatment was augmented by between-session text messaging and online community support.

SUMMARY:
This is a naturalistic, observational study of individuals with obsessive-compulsive disorder who were treated with exposure and response prevention via video teletherapy, augmented with between-session support with text messaging and an online community forum.

ELIGIBILITY:
Inclusion Criteria:

* obsessive-compulsive disorder

Exclusion Criteria:

* none

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a naturalistic sample of children, adolescents, and adults with obsessive-compulsive disorder (OCD) who sought treatment for OCD from NOCD, LLC, a digital behavioral health company.
Sampling Method: Non-Probability Sample
Enrollment: 2069 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-11-08 (Actual); Study Completion 2020-11-08 (Actual)

PRIMARY OUTCOMES:
Dimensional Obsessive-Compulsive Scale | change from pre-treatment to post-treatment (after 11 weeks)
  self-rated psychometric instrument to measure symptom severity of multiple OCD subtypes

SECONDARY OUTCOMES:
Diagnostic Interview for Anxiety, Mood, and OCD and Related Neuropsychiatric Disorders (DIAMOND) OCD severity scale | pre-treatment, after 4 weeks, and post-treatment (after 11 weeks)
  clinician-rated psychometric instrument to measure overall OCD symptom severity
Depression Anxiety and Stress Scale (DASS-21) | pre-treatment, after 4 weeks, and post-treatment (after 11 weeks)
  self-rated psychometric instrument to measure depression, anxiety, and stress
Quality of Life Enjoyment and Satisfaction Questionnaire -- Short Form (QLES-Q) | pre-treatment, after 4 weeks, and post-treatment (after 11 weeks)
  self-rated psychometric instrument to measure quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Nocd, Llc, Chicago, Illinois, United States